CLINICAL TRIAL: NCT06573489
Title: Minimum Effective Dose and Maintenance Effectiveness of Fospropofol for General Anesthesia Induction in Adult Laparoscopic Abdominal Surgery: A Randomized, Single-Blind, Clinical Study
Brief Title: Efficacy and Safety of Fospropofol in Adult Laparoscopic Surgery: A Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hui Xu (Other)
Responsible Party: Sponsor-Investigator, Hui Xu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202405048
Record Dates: First submitted 2024-08-13; First posted 2024-08-27 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Drug Safety
Keywords: Fospropofol; Efficacy and Safety
MeSH Terms: interventions — fospropofol; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fospropofol group (Experimental): patients in the fospropofol group received propofol phosphate, sufentanil, and rocuronium.
  Interventions: Drug: Fospropofol
- Propofol group (Active Comparator): patients in the propofol group received propofol, sufentanil, and rocuronium.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fospropofol — Use fospropofol for general anesthesia maintenance
  Other Names: fospropofol disodium
  Arms: Fospropofol group
Drug: Propofol — Use propofol for general anesthesia maintenance
  Other Names: Diprivan propofol
  Arms: Propofol group

SUMMARY:
This protocol is a clinical study of fospropofol disodium for general anesthesia in adults undergoing laparoscope-assisted abdominal surgery. The study has three main objectives: First, to explore the use of propofol disodium as the lowest effective dose for induction of general anesthesia; Secondly, to evaluate the efficacy and safety of fospropofol disodium in the maintenance phase of general anesthesia, and to determine its effective dose range; Finally, the effects of fospropofol disodium on Bispectral Index during induction, maintenance and recovery were studied, and compared with propofol to understand its characteristic changes. The randomized, single-blind, controlled design of the study, with an expected enrollment of 373 patients, was designed to achieve its objectives through a three-phase trial design to provide important clinical information about the safety and efficacy of the use of propofol disodium.

DETAILED DESCRIPTION:
1. To explore the lowest effective dose of fospropofol disodium for general anesthesia induction in adult laparoscopic abdominal surgery
2. Observation on efficacy, safety and effective dose range of propofol disodium for general anesthesia maintenance in adult laparoscopic abdominal surgery
3. To study the changes of Bispectral Index in the brain of patients treated with propofol during induction, maintenance and recovery of general anesthesia during laparoscopic abdominal surgery in adults, and to compare with BIS（Bispectral Index） monitoring under propofol, and to study the characteristic changes of BIS（Bispectral Index） waveform in patients treated with propofol disodium.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age (18-65 years old)
2. ASA（American Society of Anesthesiologists）grade I~II
3. The estimated operation time is more than 3h, and laparoscopic abdominal surgery under general anesthesia is planned
4. BMI value 18-30kg /m2
5. Voluntary signing of informed consent

Exclusion Criteria:

1. Those who have contraindications to general anesthesia or have a history of anesthesia accidents;
2. Patients with craniocerebral loss, intracranial hypertension, stroke, unstable angina pectoris, myocardial infarction;
3. Respiratory insufficiency, obstructive pulmonary disease, presence of a difficult airway, or determination of tracheal intubation difficulty (modified Markov score level III or IV)
4. uncontrolled diabetes or high blood pressure;
5. A history of drug use, alcoholism or drug dependence;
6. Abuse or long-term use of narcotic, sedative and analgesic drugs;
7. Those who are known or suspected to be allergic to or contraindicated by the process administration of various components or protocols of the study drug (sufentanil citrate injection, propofol medium/long chain fat milk, remifentanil hydrochloride for injection, and propofol disodium for injection);
8. People with a history of mental illness;
9. Participants in any drug clinical trial within 1 month before screening;
10. Pregnant and lactating women; The reluctance of fertile women or men to use contraception throughout the trial; Subjects (including male subjects) who plan to become pregnant within 3 months after the trial;
11. Subjects who have any other factors deemed unsuitable by the investigator for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative hypotension | From the beginning to the end of surgery
  Incidence of hypotension throughout perioperative period
Incidence of injection pain | During induction of anesthesia
  Incidence of perceived injection pain during anesthesia induction

SECONDARY OUTCOMES:
Glomerular filtration rate | First day after surgery
  The patients' glomerular filtration rate
Eeg dual frequency exponential waveform | From the beginning to the end of surgery
  Eeg dual frequency index waveform during operation
Urea nitrogen | First day after surgery
  Blood level of urea nitrogen
Creatinine | First day after surgery
  Blood level of creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Tao Hong, Master, Study Director — Tongji Hospital, Tongji Medical College, Huazhong University of Scien
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinis-Oliveira RJ. Metabolic Profiles of Propofol and Fospropofol: Clinical and Forensic Interpretative Aspects. Biomed Res Int. 2018 May 24;2018:6852857. doi: 10.1155/2018/6852857. eCollection 2018. PMID 29992157
- [Result] Patwardhan A, Edelmayer R, Annabi E, Price T, Malan P, Dussor G. Receptor specificity defines algogenic properties of propofol and fospropofol. Anesth Analg. 2012 Oct;115(4):837-40. doi: 10.1213/ANE.0b013e318258b9db. Epub 2012 May 14. PMID 22584560